CLINICAL TRIAL: NCT03499639
Title: Efficacy and Safety of Ombitasvir/ Paritaprevir / Ritonavir Plus Ribavirin in Management HCV Genotype 4 and End-stage Kidney Disease With or Without Hemodialysis (An Open Label- Multicenter Prospective Study)
Brief Title: Ombitasvir/ Paritaprevir / Ritonavir Plus Ribavirin in Management HCV and End-stage Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: Sohag University (Other); South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelsabour Mekky, Ass. Professor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 17100240
Record Dates: First submitted 2018-04-05; First posted 2018-04-17 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: End-stage Renal Disease; HCV Coinfection
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — ombitasvir; paritaprevir; Ritonavir; Ribavirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with HCV and ESKD (Other): Ombitasvir / Paritaprevir / Ritonavir/Ribavirin Oral Tablet
  Interventions: Drug: Ombitasvir / Paritaprevir / Ritonavir /Ribavirin Oral Tablet

INTERVENTIONS:
Drug: Ombitasvir / Paritaprevir / Ritonavir /Ribavirin Oral Tablet — * Patients with eGFR between 59-30ml/min: a co-formula of ombitasvir (OBV; 25mg)/ paritaprevir (PTV; 150mg)/ ritonavir (r; 100mg) (OBV/PTV/r) once-daily plus ribavirin (RIB) was given for 12 weeks. Dose adjustment of RIB was made as follow: If eGFR was 30-59 ml/min, an alternating dosing of 200 mg and 400 mg daily; if eGFR 15-30 ml/min, dosing was 200 mg once daily.
  * Patients on hemodialysis: a co-formula of OBV/PTV/r (25/150/100mg) once-daily plus RIB 200 mg 3 times/week, only in the days that they have their hemodialysis settings, 4 hours before the hemodialysis setting for 12 weeks.

SUMMARY:
Management of patients with hepatitis C virus (HCV) related liver disease with concomitant co-morbidity was challenging, especially in the period before the era of new direct-acting antiviral (DAA) agents. With the introduction of DAAs protocols, the therapeutic options were expanded to endorse many patients that were previously assigned as difficult-to-treat population. Different situations were encountered with co-infection with HCV such as chronic kidney disease (CKD) with its spectrum from mild forms to the end-stage kidney disease (ESKD), patients on hemodialysis (HD), and in post-renal transplant settings. Till now, pooled data about the safety and efficacy of different DAAs regimens in different renal situations are still under evaluation, especially in Egypt, where HCV genotype 4 the most dominating genotype. In Egypt, there were two adopted protocols for patients with HCV and CKD; the sofosbuvir-based combinations and the ombitasvir, paritaprevir, and ritonavir plus ribavirin-based combination. Sofosbuvir was proved to be contraindicated in patients with end-stage renal diseases as its elimination based mainly on renal route that may affect its bioavailability. On the other hand, ombitasvir, paritaprevir, and ritonavir plus ribavirin regimen was proved to be a well-tolerated protocol in non-cirrhotic patients with CKD.

DETAILED DESCRIPTION:
Introduction Management of patients with hepatitis C virus (HCV) related liver disease with concomitant co-morbidity was challenging, especially in the period before the era of new direct-acting antiviral (DAA) agents. With the introduction of DAAs protocols, the therapeutic options were expanded to endorse many patients that were previously assigned as difficult-to-treat population [ ]. Different situations were encountered with co-infection with HCV such as chronic kidney disease (CKD) with its spectrum from mild forms to the end-stage kidney disease (ESKD), patients on hemodialysis (HD), and in post-renal transplant settings [ , ]. Till now, pooled data about the safety and efficacy of different DAAs regimens in different renal situations are still under evaluation [ ], especially in Egypt, where HCV genotype 4 the most dominating genotype [ ]. In Egypt, there were two adopted protocols for patients with HCV and CKD; the sofosbuvir-based combinations and the ombitasvir, paritaprevir, and ritonavir plus ribavirin-based combination [5, ]. Sofosbuvir was proved to be contraindicated in patients with end-stage renal diseases as its elimination based mainly on renal route that may affect its bioavailability [ ]. On the other hand, ombitasvir, paritaprevir, and ritonavir plus ribavirin regimen was proved to be a well-tolerated protocol in non-cirrhotic patients with CKD [6, ].

Aim Therefore, we herein, tried to evaluate a real-life practice to evaluate the efficacy and safety of ombitasvir, paritaprevir, and ritonavir plus ribavirin regimen in patients with ESKD, with or without hemodialysis in Egyptian based multicenter cohort.

Patients and Methods

Patients' recruitment:

Starting from July 2017, a prospective multicenter cohort study was designed to enroll all consecutive patients presented at the Viral Hepatitis Management Outpatient Clinic at Assiut University Hospital, South Valley University Hospital, Sohag University Hospital, Egypt, with proven CHC genotype 4 and concomitant ESKD with or without hemodialysis.

Enrolled patients were 18 years old or more, naive to HCV treatment, HCV genotype 4, and compensated liver disease. Patients with combined HCV/HBV co-infection, hepatocellular carcinoma (HCC), decompensated liver cirrhosis (Child-Pugh score above 6), and non-genotype 4 were excluded.

Study definitions

* ESKD was based on estimated glomerular filtration rate (eGFR) that calculated by the Cockroft-Gault equation [ , ].
* Two sets of patients: ESKD-group; eGFR less than between 59-30 ml/min without hemodialysis and HD-group; eGFR less than 30 ml/min with or without hemodialysis
* HCV Treatment Response: sustained virologic response was defined as HCV RNA under the detection limit at week 12 after the end of treatment (SVR12), non-responder was defined as a detectable viremia at week 12, and relapse was defined as re-appearance of HCV viremia during follow up after being undetectable at week 12 [ ].

Study methods and follow up protocol

* Liver disease-status was assessed before therapy by Child-Turcotte Pugh (CTP) score [ ] and liver stiffness score measurements by Fibroscan® (EchoSens, Paris, France) in kilopascals (kPa) according to the manufacturer's instructions (score less than 7.4 kPa equal to F0-F2, 9.5-12.4 kPa equal to F3, and 14.5 kPa or greater equal to F4 on METAVIR pathologic scoring system) [ , ].
* HCV genotype assessment by direct sequencing of the 50 untranslated region (50UTR), using RT-PCR-based assay (AmpliSens HCV-genotype-FRT PCR kit).
* HCV RNA was measured using the Roche COBAS Taq Man HCV assay version 2.0 (lower limit of detection 15 IU/mL).
* In all patients, hematologic (hemoglobin level) liver (CTP score parameters), renal (eGFR), and virologic (HCV-RNA viremia), and the co-medications such as immunosuppressive drugs (doses and levels), were evaluated at base-line (week0), at weeks 4, 12 during therapy, and week 24 after.

HCV Medications & protocols (Figure 1)[according to the National Committee for Control of Viral Hepatitis (NCCVH)]

* Patients with eGFR between 59-30ml/min: a co-formula of ombitasvir (OBV; 25mg)/ paritaprevir (PTV; 150mg)/ ritonavir (r; 100mg) (OBV/PTV/r) once-daily plus ribavirin (RIB) was given for 12 weeks. Dose adjustment of RIB was made as follow: If eGFR was 30-59 ml/min, an alternating dosing of 200 mg and 400 mg daily; if eGFR 15-30 ml/min, dosing was 200 mg once daily.
* Patients on hemodialysis: a co-formula of OBV/PTV/r (25/150/100mg) once-daily plus RIB 200 mg 3 times/week, only in the days that they have their hemodialysis settings, 4 hours before the hemodialysis setting for 12 weeks.

Study outcome measures & endpoints The primary endpoint was the achievement of SVR at week 12 (SVR12) post-treatment. The potential adverse events were evaluated in each visit for the development of adverse events or any significant interactions.

Statistical analysis and ethical considerations Frequencies, percentages, and means were used, as appropriate, for descriptive analysis. Chi Square test was used to compare parametric qualitative data, while Mann-Whitney test was used to compare non-parametric qualitative data and fisher exact test used to compare non-parametric qualitative data. Statistical analysis was conducted by SPSS (V.19, SPSS Inc.; Chicago, IL, USA). A p-value < 0.05 was considered significant. The study was approved by the local Ethical Committee.

ELIGIBILITY:
Inclusion Criteria:

* patients were 18 years old or more,
* naive to HCV treatment,
* HCV genotype 4,
* compensated liver disease.

Exclusion Criteria:

* Patients with combined HCV/HBV co-infection
* hepatocellular carcinoma (HCC)
* decompensated liver cirrhosis (Child-Pugh score above 6)
* non-genotype 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was the achievement of SVR at week 12 (SVR12) post-treatment. | 6 months

SECONDARY OUTCOMES:
The potential adverse events were evaluated in each visit for the development of adverse events or any significant interactions. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Mekky, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hopsital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
share through publishing a scientific paper